CLINICAL TRIAL: NCT00852605
Title: A Randomized Clinical Trial on the Use of Early Intermittent Non-Invasive Ventilation in Patients Suffering From Acute Lung Injury After Allogeneic Transplantation
Brief Title: Acute Lung Injury After Allogeneic Transplantation - Diagnosis and Early Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Masking: None
Other Study IDs: NIV2001
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Acute Lung Injury
Keywords: Acute Lung Injury after allogeneic transplantation
MeSH Terms: conditions — Acute Lung Injury

ARMS (2):
- Oxygen (No Intervention): Conventional Treatment including Oxygen-support
- NIV (Experimental): Conventional Treatment plus intermittent Non-Invasive-Ventilation
  Interventions: Other: Intermittent Non-Invasive Ventilation

INTERVENTIONS:
Other: Intermittent Non-Invasive Ventilation
  Arms: NIV

SUMMARY:
Acute lung injury (ALI) is an early complication after allogeneic transplantation causing significant mortality and morbidity. Little is known on early markers and treatment of this complication. Recent data (Hilbert et al.) suggested a beneficial effect of Non-Invasive-Ventilation in ALI-patients immunosuppressed because a many different reasons including stem-cell transplantation.

The investigators study is designed to evaluate early markers of ALI after allogeneic transplantation. In case ALI is documented patients are randomized to either conventional therapy (oxygen-support) or conventional therapy plus intermittent Non-Invasive Ventilation. The hypothesis is that Non-Invasive Ventilation improves outcome of ALI after allogeneic transplantation.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing allogeneic transplantation presenting with at least two of the following criteria

* Respiratory rate >25 / min
* Oxygenation Index <300
* Continuous oxygen-saturation <92% whilst breathing room air

Exclusion Criteria:

* Indication for Emergency intubation
* Hemodynamic instability
* Left ventricular failure
* GCS <8
* No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2001-12; Primary Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Illmer Thomas, Ph D, Principal Investigator — Medizinische Klinik I - Universitätsklinikum Carl-Gustav-Carus Dresden